CLINICAL TRIAL: NCT01080599
Title: Comparison of the Success Rate of Two Approaches for Obturator Nerve Block in TURB (Conventional Pubic Approach [Labat Technique] and Inguinal Approach)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Hae Keum Kil/Professor, Yonsei University, College of Medicine
Allocation: Randomized | Model: Parallel
Other Study IDs: 4-2009-0137
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Nerve Block
Keywords: obturator nerve block in TURB

ARMS (2):
- conventional pubic approach (Experimental)
  Interventions: Procedure: obturator nerve block
- inguinal approach (Experimental)
  Interventions: Procedure: obturator nerve block

INTERVENTIONS:
Procedure: obturator nerve block

SUMMARY:
The purpose of this study is to compare the success rate of two approaches for obturator nerve block in TURB (conventional pubic approach [Labat technique] and inguinal approach.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergoing transurethral resection of bladder tumor during combined spinal anesthesia and obturator nerve block were included in the clinical study

Exclusion Criteria:

* Patients with advanced cardiac and respiratory insufficiency
* Allergy to local anesthetics
* Preexisting neurologic deficits
* Prior operation involving the hip and the inguinal region and bleeding tendency were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Assessment of obturator sign during using nerve stimulator and operation